CLINICAL TRIAL: NCT00655382
Title: Dynamic MRI Evaluation Post op STARR Procedure
Brief Title: Dynamic MRI Evaluation Post Operative Stapled Trans Anal Rectal Resection (STARR) Procedure
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Paul D. Pettit, M.D., Mayo Clinic
Other Study IDs: 06-004724
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2010-05-21 (Estimated); Status verified 2010-05

CONDITIONS: Obstructive Defecation Syndrome; Outlet Obstruction
Keywords: dynamic pelvic mri; dynamic mri; STARR procedure; STARR; ODS; obstructive defecation syndrome; outlet obstruction; obstructed defecation; stapled trans anal rectal resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to assess the effects of the Stapled Trans Anal Rectal Resection (STARR) procedure for patients with obstructive defecation syndrome. This involves a dynamic pelvic MRI and obstructive defecation score (ODS) at 6 month post STARR procedure.

DETAILED DESCRIPTION:
The use of dynamic pelvic MRI has greatly impacted our preoperative evaluation of pelvic floor disorders, both anatomically and functionally. The STARR procedure is a new approved procedure for patients with obstructive defecation, who have failed conservative therapy of medications and aggressive pelvic floor retraining. Most patients have also been screened for colonic transit problems. The traditional study for evaluating these patients was defecating proctograms. With the advent of the dynamic pelvic MRI, we are now beginning to understand the interaction of the entire pelvic structure in the complex act of defecation. This study is providing us a different view of the pelvic structures to better understand the pathophysiology of this disorder. The defecating proctogram, though informative in certain cases, lacks information outside the rectum. We wish to evaluate and compare our preoperative dynamic pelvic MRI with a six month dynamic pelvic MRI in 10 patients. We also will compare pre and post op obstructive defecation scores (ODS). We expect this small sample to direct us to a much more pointed evaluation of this disorder.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to have a follow-up with a dynamic pelvic MRI and complete an obstructive defecation score (ODS) at 6 month post STARR procedure at Mayo Clinic - Jacksonville

Exclusion Criteria:

* Patients with medical devices/implants or who cannot have follow-up dynamic pelvic MRI

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had STARR procedure performed at Mayo Clinic - Jacksonville
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2007-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul D. Pettit, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States